CLINICAL TRIAL: NCT03963726
Title: Clinical Efficacy of Stereotactic Radiotherapy and Microwave Ablation for Liver Metastases From Colorectal Cancer: a Prospective Multicenter Cohort Study
Brief Title: Clinical Efficacy of Stereotactic Radiotherapy and Microwave Ablation for Liver Metastases From Colorectal Cancer.
Acronym: Ckvsmalm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beijing 302 Hospital (Other); Tengzhou Central People's Hospital (Other Government); Guangxi Ruikang Hospital (Other); Hunan Aerospace Hospital (Unknown); Beijing Ditan Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BYSY-CKMA-LM
Record Dates: First submitted 2019-05-21; First posted 2019-05-28 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-05

CONDITIONS: Radiotherapy; Microwave Ablation; Liver Metastases; Colorectal Cancer
Keywords: Radiotherapy; microwave ablation; Liver Metastases; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: non-randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Stereotactic radiotherapy (Experimental): In this study, the liver metastases were treated with Cyberknife stereotactic radiotherapy.Using multimodal image fusion to outline the target area.According to the volume, location, organ function and other factors, the dosage of radiotherapy was determined. The range of BED value of radiotherapy was 90-120 when the distance between the tumor and gastrointestinal tract was more than 5 mm (alpha/beta=10) and 70-90 when the distance between the tumor and gastrointestinal tract was less than 5 mm (alpha/beta=10).
  Interventions: Radiation: stereotactic radiotherapy
- Microwave ablation therapy (Experimental): In this study, 3D printing template was used to assist microwave ablation.For those whose lesions are directly smaller than 5.0cm, the ablation time is about 10 min and 15 min, and the ablation time is more than 15min in patients larger than 5.0cm.
  Interventions: Other: microwave alabation

INTERVENTIONS:
Radiation: stereotactic radiotherapy — The liver metastases were treated with Cyberknife stereotactic radiotherapy.Using multimodal image fusion to outline the target area.According to the volume, location, organ function and other factors, the dosage of radiotherapy was determined. The range of BED value of radiotherapy was 90-120 when the distance between the tumor and gastrointestinal tract was more than 5 mm (alpha/beta=10) and 70-90 when the distance between the tumor and gastrointestinal tract was less than 5 mm (alpha/beta=10).
  Arms: Stereotactic radiotherapy
Other: microwave alabation — The colorectal cancer patients with liver metastases will receive microwave ablation.3D printing template was used to assist microwave ablation.For those whose lesions are directly smaller than 5.0cm, the ablation time is about 10 min and 15 min, and the ablation time is more than 15min in patients larger than 5.0cm.
  Arms: Microwave ablation therapy

SUMMARY:
Data of 100 colorectal cancer patients with liver metastases who received stereotactic radiotherapy of Cyberknife or microwave ablation in the multicenter of the research group from June 2019 to May 2021 were collected, as well as follow-up data.To evaluate the clinical efficacy of stereotactic radiotherapy and microwave ablation in liver metastases.In addition, the local control rate and side effects of stereotactic radiotherapy and microwave ablation in the treatment of liver metastases were explored, and the efficacy and safety of different doses of stereotactic radiotherapy were determined.

DETAILED DESCRIPTION:
In the study，data of 100 colorectal cancer patients with liver metastases who received Cyberknife stereotactic radiotherapy or microwave ablation in the multi-center of the research group from June 2019 to May 2021 were collected, as well as follow-up data.

1. Radiation: Stereotactic Radiotherapy 1.1 Equipment: Accuray VSI Cyberknife stereotactic radiotherapy platform, simulated positioning CT machine, MR, positron emission computed tomography PET-CT, vacuum pad.

   1.2 Radiotherapy localization: CT, MRI and PETCT were used to simulate localization.

   1.3 Relevant Definitions of Tumor Targets CT, MRI, PET-CT fusion, combined with MRI location and PET-CT location image for sketching.

   To delineate target areas and organs at risk. GTV: Combining localization and fusion images to delineate the tumors seen PTV = GTV + 0-10mm Dangerous organs: The stomach, duodenum, jejunum, ileum, colon, spinal cord and esophagus were delineated on the base sequence of CT plain scan.

   The target area should be approved by at least one physician in charge or by a physician in charge.

   1.4 Target volume radiation dose: According to the volume, location, organ function and other factors, the dosage of radiotherapy was determined. The range of BED value of radiotherapy was 90-120 when the distance between the tumor and gastrointestinal tract was more than 5 mm (alpha/beta=10) and 70-90 when the distance between the tumor and gastrointestinal tract was less than 5 mm (alpha/beta=10).

   1.5 Normal Tissue Limit: Reference to TG101 Report
2. Microwave ablation 2.1 Preoperative positioning and planning: 2.1.1 Determine the fixing device: generally choose vacuum pad to fix 2.1.2 Choosing the right position: The principle is to choose the position that is easy to operate, taking into account the comfort and tolerance of patients.

2.1.3 CT scan 2.1.4 The range of tumors was determined by CT images. In principle, at the maximum level, the skin points corresponding to the vertical center of the tumor are the marker points of the locating needle. At the same time, the center of the tumor was taken as the origin point, and the longitudinal and transverse cross lines were drawn on the patient's body surface. Roughly delineate the range of tumors according to CT in body surface 2.2 Surgery and intraoperative optimization 2.2.1 Posture reduction and fixation of patients 2.2.2 Oxygen inhalation, ECG and blood pressure monitoring 2.2.3 Installation of 3D Printing Planar Coordinate Template Fixer 2.2.4 Routine disinfection, cave towel laying, local infiltration anesthesia, fixing 3D printing plane coordinate template according to the range of tumors determined by physical examination and preoperative plan, and adjusting the direction of plane template by protractor.

2.2.5 Puncture locating needle and puncture assistant fixing needle in 4 directions of tumor margin.

2.2.6The real-time CT 2.5mm image was imported into the navigation system, the puncture needle was marked, the puncture needle was simulated, and the resolution of the template was adjusted accurately.

2.2.7 Enhanced CT scan to determine the position and angle of template and pin accurately 2.2.8 Layer by layer puncture according to preoperative plan 2.2.9 After inserting the ablation antenna to the reserved position, scan CT again to confirm whether the puncture needle has reached the planned position. 2.2.10 Complete ablation of tumors as planned.

2.3Postoperative observation 2.3.1 With the assistance of the staff in the hospital, they will be transported back to the ward by flat car with their families.

2.3.2 Re-measurement of blood pressure and heart rate 2.3.3Observe whether there is bleeding or exudation at the puncture point after operation, and give hemostasis and pain relief if necessary.

To evaluate the clinical efficacy of stereotactic radiotherapy and microwave ablation in liver metastases after these treatment.In addition, the local control rate and side effects of stereotactic radiotherapy and microwave ablation in the treatment of liver metastases were explored, and the efficacy and safety of different doses of stereotactic radiotherapy were determined.

ELIGIBILITY:
Inclusion Criteria:

* The age was 18 to 80 years old.
* It was confirmed by pathology that the liver metastasis of colorectal cancer was less than or equal to 3 lesions, each lesion was less than 3 cm, and there was no invasion of vascular tumor thrombus and adjacent organs according to the discussion of MDT.
* The preoperative imaging evaluation of iatrogenic or / and personal factors can realize microwave ablation or radiosurgery SBRT to require.
* The primary lesion has been treated radical and has no evidence of recurrence, and there is no metastasis outside the liver.
* The physical status score of ECOG : 0 ≥ 1 or more than 60 KPS.
* Predicted survival time was more than 3 months.
* The main organ function can tolerate stereotactic radiotherapy / microwave ablation, liver function child-pugh A or B, no severe hypertension, diabetes and heart disease. That is, within 14 days of random examination, the relevant test indexes meet the following requirements:

  1. blood routine examination: i. Hemoglobin was more than 90 g /L (no blood transfusion); ii. Neutrophil count was more than 1.5x109/L; iii platelet count was more than 100x109/ L;
  2. biochemical examination: i. total cholerythrin-1.5-ultraln (upper limit of normal); ii. Blood-valley-pyruvic transaminase (ALT) or blood-glutamic-aspartate aminotransferase (AST), 2.5-hulled; iii. The clearance of endophytic muscle was 60 ml/ min (ckroft-gault formula);
  3. cardiac Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) was more than 50%;
  4. blood glucose control was less than 7.2 mmol/ L, non-fasting blood glucose was less than 10 mmol/L, and glycosylated hemoglobin was less than 7%.
* Sign informed consent form.
* Good compliance, family agreed to cooperate with follow-up.

Exclusion Criteria:

* Patients who are being treated with drugs and whose liver metastases are stable or relieved, and who have participated in clinical trials of other drugs within four weeks;
* There was a history of bleeding, and any serious bleeding events of 3 degrees or more in ctcae 5.0 occurred within 4 weeks before screening.
* Patients with known central nervous system metastasis or history of central nervous system metastasis before screening. For patients with suspected central nervous system metastasis, CT or MRI examination must be performed within 14 days before randomization to exclude central nervous system metastasis.
* Patients with high blood pressure and single step-down medications were not able to obtain good control (systolic blood pressure was more than 140 mmHg, diastolic blood pressure was more than 90 mmHg); patients with a history of unstable angina; a new diagnosis within 3 months before screening was an event of myocardial infarction within 6 months before or after screening; Arrhythmias (including QTCF: male,450 ms, female, 470ms) require long-term use of anti-arrhythmic drugs and the New York Heart Association rating of grade ii cardiac insufficiency;
* Long-term unhealed wounds or incomplete fractures,
* Imaging showed that the tumor had invaded the perivascular area of important vessels or was judged by researchers that the tumor was highly likely to invade important blood vessels during treatment, resulting in fatal massive bleeding.
* Patients with abnormal coagulation function and bleeding tendency (14 days before randomization must be satisfied:INR is within the normal range without anticoagulant); Patients treated with anticoagulant or vitamin k antagonists such as warfarin, heparin or its analogues; Low dose warfarin (1mg oral, once a day) or low dose aspirin (not exceeding 100 mg); per day) is allowed for prophylactic purposes on the premise that the international standardized ratio of prothrombin time (INR) was less than 1.5;
* Hyperarteriovenous thrombosis occurred within 6 months before screening, such as cerebrovascular accidents (including temporary ischemic seizures), Deep venous thrombosis (except where venous thrombosis caused by intravenous catheterization after pre-chemotherapy has been cured by researchers) and pulmonary embolism, etc.
* There was abnormal thyroid function in the past, and even in the case of drug treatment, thyroid function could not be maintained within the normal range;
* Having a history of psychotropic substance abuse and unable to give up or have mental disorders.
* Radiotherapy for abdominal tumors has been carried out in the past.
* Have a history of immunodeficiency, or suffer from other acquired, congenital immunodeficiency diseases, or have a history of organ transplantation.
* According to the researchers' judgment, there are serious diseases that endanger the safety of patients or affect the completion of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-06-03 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Local control rate | 3 years after the treatment
  Local control refers to the fact that the tumor is not enlarged on imaging, but if the tumor is not enlarged, the patients with aggravated symptoms after treatment are not included in the local control range.
Objective response rate | 1 years after the treatment
  The proportion of patients whose tumors have shrunk to a certain extent and maintained for a certain period of time, including CR + PR cases
Disease control rate | 3 years after the treatment
  After treatment, the number of cases with remission and stable lesions accounted for the percentage of the total number of assessable cases
PFS | 3 years after the treatment
  The time interval of disease progression since the date of diagnosis

SECONDARY OUTCOMES:
Overall survival | 3 years after the treatment
  The time from enrollment to death from any cause
Side effects | 1 years after the treatment
  Harmful reactions unrelated to the purpose of treatment occur in the course of the treatment of a disease
Quality of life score of tumor patients(0-60) | 3 years after the treatment
  Common methods for evaluating the quality of life of patients:The full score of quality of life is 60, the worst is < 20, the worse is 21-30, the average is 31-40, the better is 41-50, and the good is 51-60.

CONTACTS AND LOCATIONS:
Overall Officials: Junjie U Wang, MD, Study Chair — Peking University Third Hospital; Fei U Xu, M Med, Study Director — Peking University Third Hospital; Xuezhang Duan, MD, Principal Investigator — Beijing 302 Hospital; Kaixian Zhang, MD, Principal Investigator — Tengzhou Central People's Hospital; Wei Li, MD, Principal Investigator — Beijing Ditan Hospital; Hui Xie, MD, Principal Investigator — Beijing 302 Hospital; Zuping Lian, MD, Principal Investigator — Guangxi Ruikang Hospital; Xian Xu, M Med, Principal Investigator — Hunan Aerospace Hospital; Fuxin Guo, MD, Principal Investigator — Peking University Third Hospital; Jing Sun, M Med, Principal Investigator — Beijing 302 Hospital
Locations (6):
- China (6):
  - Beijing Ditan Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The fifth medical center of PLA general hospital, Beijing, Beijing Municipality
  - Guangxi ruikang hospital, Nanning, Guangxi
  - Hunan Aerospace Hospital, Changsha, Hunan
  - Tengzhou Central People's Hospital, Tengzhou, Shandong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yuan ZY, Meng MB, Liu CL, Wang HH, Jiang C, Song YC, Zhuang HQ, Yang D, Wang JS, Wei W, Li FT, Zhao LJ, Wang P. Stereotactic body radiation therapy using the CyberKnife((R)) system for patients with liver metastases. Onco Targets Ther. 2014 Jun 12;7:915-23. doi: 10.2147/OTT.S58409. eCollection 2014. PMID 24959080
- [Background] Mihara K, Kaihara M, Sunahori S, Yamashiro N, Nishiya S, Ito Y, Funakoshi K, Egawa T, Tsukamoto N, Nagashima A. [Stereotactic Body Radiotherapy with CyberKnife(R)for Liver Metastases from Colorectal Cancer]. Gan To Kagaku Ryoho. 2015 Oct;42(10):1262-4. Japanese. PMID 26489566
- [Background] Kress MS, Collins BT, Collins SP, Dritschilo A, Gagnon G, Unger K. Stereotactic body radiation therapy for liver metastases from colorectal cancer: analysis of safety, feasibility, and early outcomes. Front Oncol. 2012 Feb 2;2:8. doi: 10.3389/fonc.2012.00008. eCollection 2012. PMID 22649775
- [Background] Dewas S, Bibault JE, Mirabel X, Fumagalli I, Kramar A, Jarraya H, Lacornerie T, Dewas-Vautravers C, Lartigau E. Prognostic factors affecting local control of hepatic tumors treated by Stereotactic Body Radiation Therapy. Radiat Oncol. 2012 Oct 10;7:166. doi: 10.1186/1748-717X-7-166. PMID 23050794
- [Background] Herfarth KK, Debus J, Wannenmacher M. Stereotactic radiation therapy of liver metastases: update of the initial phase-I/II trial. Front Radiat Ther Oncol. 2004;38:100-5. doi: 10.1159/000078271. No abstract available. PMID 15458194
- [Background] Mendez Romero A, Wunderink W, Hussain SM, De Pooter JA, Heijmen BJ, Nowak PC, Nuyttens JJ, Brandwijk RP, Verhoef C, Ijzermans JN, Levendag PC. Stereotactic body radiation therapy for primary and metastatic liver tumors: A single institution phase i-ii study. Acta Oncol. 2006;45(7):831-7. doi: 10.1080/02841860600897934. PMID 16982547
- [Background] Hoyer M, Roed H, Traberg Hansen A, Ohlhuis L, Petersen J, Nellemann H, Kiil Berthelsen A, Grau C, Aage Engelholm S, Von der Maase H. Phase II study on stereotactic body radiotherapy of colorectal metastases. Acta Oncol. 2006;45(7):823-30. doi: 10.1080/02841860600904854. PMID 16982546
- [Background] Lee MT, Kim JJ, Dinniwell R, Brierley J, Lockwood G, Wong R, Cummings B, Ringash J, Tse RV, Knox JJ, Dawson LA. Phase I study of individualized stereotactic body radiotherapy of liver metastases. J Clin Oncol. 2009 Apr 1;27(10):1585-91. doi: 10.1200/JCO.2008.20.0600. Epub 2009 Mar 2. PMID 19255313
- [Background] Lanciano R, Lamond J, Yang J, Feng J, Arrigo S, Good M, Brady L. Stereotactic body radiation therapy for patients with heavily pretreated liver metastases and liver tumors. Front Oncol. 2012 Mar 9;2:23. doi: 10.3389/fonc.2012.00023. eCollection 2012. PMID 22645716
- [Background] Ambrosino G, Polistina F, Costantin G, Francescon P, Guglielmi R, Zanco P, Casamassima F, Febbraro A, Gerunda G, Lumachi F. Image-guided robotic stereotactic radiosurgery for unresectable liver metastases: preliminary results. Anticancer Res. 2009 Aug;29(8):3381-4. PMID 19661360
- [Background] Rusthoven KE, Kavanagh BD, Cardenes H, Stieber VW, Burri SH, Feigenberg SJ, Chidel MA, Pugh TJ, Franklin W, Kane M, Gaspar LE, Schefter TE. Multi-institutional phase I/II trial of stereotactic body radiation therapy for liver metastases. J Clin Oncol. 2009 Apr 1;27(10):1572-8. doi: 10.1200/JCO.2008.19.6329. Epub 2009 Mar 2. PMID 19255321
- [Background] Katz AW, Carey-Sampson M, Muhs AG, Milano MT, Schell MC, Okunieff P. Hypofractionated stereotactic body radiation therapy (SBRT) for limited hepatic metastases. Int J Radiat Oncol Biol Phys. 2007 Mar 1;67(3):793-8. doi: 10.1016/j.ijrobp.2006.10.025. Epub 2006 Dec 29. PMID 17197128
- [Background] Yamashita H, Onishi H, Matsumoto Y, Murakami N, Matsuo Y, Nomiya T, Nakagawa K; Japanese Radiological Society multi-institutional SBRT study group (JRS-SBRTSG). Local effect of stereotactic body radiotherapy for primary and metastatic liver tumors in 130 Japanese patients. Radiat Oncol. 2014 May 10;9:112. doi: 10.1186/1748-717X-9-112. PMID 24886477
- [Background] Benedict SH, Yenice KM, Followill D, Galvin JM, Hinson W, Kavanagh B, Keall P, Lovelock M, Meeks S, Papiez L, Purdie T, Sadagopan R, Schell MC, Salter B, Schlesinger DJ, Shiu AS, Solberg T, Song DY, Stieber V, Timmerman R, Tome WA, Verellen D, Wang L, Yin FF. Stereotactic body radiation therapy: the report of AAPM Task Group 101. Med Phys. 2010 Aug;37(8):4078-101. doi: 10.1118/1.3438081. PMID 20879569
- [Background] Groeschl RT, Pilgrim CH, Hanna EM, Simo KA, Swan RZ, Sindram D, Martinie JB, Iannitti DA, Bloomston M, Schmidt C, Khabiri H, Shirley LA, Martin RC, Tsai S, Turaga KK, Christians KK, Rilling WS, Gamblin TC. Microwave ablation for hepatic malignancies: a multiinstitutional analysis. Ann Surg. 2014 Jun;259(6):1195-200. doi: 10.1097/SLA.0000000000000234. PMID 24096760
- [Background] Xu S, Hu K, Huang H, Yao Z, Wang Q, Yang P, Liu B, Yang Y, Chen G. [Effect of laparoscopic hepatectomy and microwave ablation for colorectal liver metastases]. Zhonghua Yi Xue Za Zhi. 2015 Oct;95(40):3289-92. Chinese. PMID 26815350